CLINICAL TRIAL: NCT05120050
Title: Clinical Evaluation of ASP Health's Automated ROSE System for Bronchoscopic Applications
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ASP Health (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ASP_LT_004
Record Dates: First submitted 2021-10-20; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Lung Diseases; Lung Cancer
Keywords: Slide deposition; Slide stainer; Automated; Pahtology
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Cytological specimens

GROUPS / COHORTS (1):
- Patients with confirmed Lung cancer
  Interventions: Device: ASP Health instrument

INTERVENTIONS:
Device: ASP Health instrument — The instrument is an integrated device with a short processing time (measured in 2 to 3 minutes) that distributes cells from limited volume samples (measured in microliters). The process involves a novel aerosolization technique that transfers liquid sample to a glass slide via a burst of air. After the sample is deposited on the glass slide, the automated system uses an integrated heating strip to heat the specimen slide. This process is similar to using a hair dryer to dry the specimen slide in the current ROSE setting. After drying the slide, the system uses series of pumps to dispense microliters of stain reagent onto the slide to stain the cells. Currently, the system is configured to perform DiffQuik staining, which is commonly used in the ROSE process. In the future, the staining capability will be broadened to include other staining processes such as Rapid PAP, H&E staining etc.

SUMMARY:
Prospective comparison of cytology slides (bronchoscopically derived fine needle aspiration samples of lymph nodes at the time of rapid intraprocedural on site evaluation) created with the ASP Health's specimen preparation system to slides made by existing conventional methods.

DETAILED DESCRIPTION:
Rapid On-Site Evaluation (ROSE) has dramatically improved patient care during Fine Needle Aspiration procedures by providing adequacy feedback to the proceduralists. In the case of endobronchial ultrasound (EBUS) procedures, the samples that are collected from the patients are reviewed to determine adequacy of samples to ensure diagnostic quality samples are being processed. If the amount of specimen is found to be adequate, the interventional pulmonologists make additional passes to collect more specimen sample. While the existing ROSE method performed by smearing the samples on the glass slide and staining the slides has dramatically improved patient outcomes, it has several challenges/drawbacks. Some of the challenges of ROSE slide preparation include: (i) high variability in sample quality, (ii) cumbersome process in the procedure room and (iii) possibility of cross contamination between samples, (iv) slow specimen preparation and staining process which leads to extended procedure time and (v) the cost of the personnel to prepare slides. The goal of this study is to conduct a trial of a novel automated sample preparation system from ASP Health that combines both the specimen deposition and staining in a compact/mobile unit. This automated system is expected to improve the workflow of the cytotechnologists and cytopathologists by ensuring reproducibility and efficiency.

ASP's sample preparation instrument: The instrument is an integrated device with a short processing time (measured in 2 to 3 minutes) that distributes cells from limited volume samples (measured in microliters). The process involves a novel aerosolization technique that transfers liquid sample to a glass slide via a burst of air. After the sample is deposited on the glass slide, the automated system uses an integrated heating strip to heat the specimen slide. This process is similar to using a hair dryer to dry the specimen slide in the current ROSE setting. After drying the slide, the system uses series of pumps to dispense microliters of stain reagent onto the slide to stain the cells. Currently, the system is configured to perform DiffQuik staining, which is commonly used in the ROSE process. In the future, the staining capability will be broadened to include other staining processes such as Rapid PAP, H&E staining etc.

The early prototype of this instrument has been successfully tested at Cleveland Clinic on residual of EBUS samples, serous body fluids, and bench top FNAs with high diagnostic concordance.

ELIGIBILITY:
Inclusion Criteria:

* Anyone who is undergoing EBUS procedure for diagnosis or staging of lung diseases.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort will be selected from patients visiting the pulmonology clinic for suspected lung lesions/diseases.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Evaluation of ASP Health's Instrument for Bronchoscopic Applications | 1 month from time of sample collection
  Confirm that ASP Health's Instrument performance is not inferior to the standard of care procedures.

SECONDARY OUTCOMES:
ASP Health's Instrument compared to standard of care | 1 week from sample collection
  ASP Health's Instrument has an improved clinical workflow compared to the standard of care procedures.